CLINICAL TRIAL: NCT02268097
Title: Comparison of Two Methods of Patellar Resurfacing in Total Knee Arthroplasty.A Prospective, Randomized, Double-blind Study
Brief Title: Comparison of Two Methods of Patellar Resurfacing in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jia-kuo yu, Peking University Third Hospital, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YJK-003
Record Dates: First submitted 2014-10-11; First posted 2014-10-20 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2014-10

CONDITIONS: Osteoarthritis
Keywords: patella; total knee arthroplasty; resection
MeSH Terms: conditions — Osteoarthritis; Patella Fracture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Freehand (Experimental): Patellar resurfacing with freehand technique:Using freehand technique for patella preparation during total knee arthroplasty.
  Interventions: Procedure: Patellar resurfacing with freehand technique
- Resection guide (Active Comparator): Patellar resurfacing with resection guide technique: Using patellar resection guide technique for patella preparation during total knee arthroplasty.
  Interventions: Procedure: Patellar resurfacing with resection guide technique

INTERVENTIONS:
Procedure: Patellar resurfacing with freehand technique — Preparing patellar resurfacing during total knee arthroplasty with freehand
  Arms: Freehand
Procedure: Patellar resurfacing with resection guide technique — Preparing patellar resurfacing during total knee arthroplasty with a resection guide
  Arms: Resection guide

SUMMARY:
The aim of this prospective, randomized study was to compare the clinical and radiological results of "free-hand" technique and "resection guide" technique for preparing patella during total knee arthroplasty.

DETAILED DESCRIPTION:
With improved surgical techniques and implant designs, patella resurfacing has been favored by increasing surgeons. When performing the resection, several principles such as restoring the original patellar thickness, avoiding over or under resection must be complied in order to achieve satisfactory outcomes.This study was conducted to compared the outcomes of two commonly adopted methods for performing patellar resection in total knee arthroplasty. One hundred patients with osteoarthritis were recruited in the clinical trial using Nexgen Legacy Posterior Stabilized-Flex prosthesis. Patients were randomized to receive "free-hand" technique and "resection guide" technique when performing patellar resection in total knee arthroplasty. Patients were evaluated preoperatively and at follow-up visits conducted at twelve months, at twenty-four months. Clinical outcome was assessed and compared with use of the visual analogue pain scale (VAS), range of motion, Knee Society Score (KSS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Short Form-36 (SF-36). Patellar alignment was assessed before surgery and at each follow-up by measuring the patellar tilt (PT) and lateral patellar displacement (PD). Prosthetic position and leg alignment were also compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of primary osteoarthritis of the knee, with Ahlbäck grade of ≥2 (symptoms persisting after conservative treatment for at least 3 months) knees with <20° varus or <15° valgus deformity patellar thickness is more than 21mm

Exclusion Criteria:

restricted motion (flexion contracture of >25°) patella alta (Insall-Salvati ratio of <0.6) history of previous knee surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2017-07-15 (Estimated); Study Completion 2017-07-15 (Estimated)

PRIMARY OUTCOMES:
Patellar tilt (PT) | 1 year
  The patellar tilt is the angle between the transverse axis of the patella and The patellar tilt is the angle between the transverse axis of the patella and the anterior intercondylar line.The PT was assessed by a blinded observer using 30° skyline radiographs.

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 1 year
  The Knee Society's Knee Scoring System (KSS) has served as a simple, objective way to measure a patient's functional ability before and after total knee arthroplasty (TKA).Scale Name:score scale range:0~100,and a higher values represent a better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 1 year
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis (OA) Index is a tested questionnaire to assess symptoms and physical functional disability in patients with OA of the knee.Scale Name:score scale range:0~100,and a lesser values represent a better outcome.
visual analogue pain scale (VAS) | 1 year
  Pain rating scales.Scale Name:score scale range:0~100,and a higher values represent a worse outcome
Short Form-36 (SF-36) | 1 year
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. A higher values represent a better outcome.
leg alignment | 1 year
  Radiographic evaluation:The measurements were made by a blinded observer, in accordance with the principles stipulated by the Knee Society, by using computer-generated data derived from the digital radiographs.
prosthetic position | 1 year
  Radiographic evaluation:The following parameters were measured: the coronal femoral component angle (α; angle between femoral shaft and transcondylar line of the femoral component); coronal tibial component angle (β; angle between the mechanical axis of the tibia and tibial base plate); sagittal femoral component angle (γ; angle of femoral component flexion); and sagittal tibial component angle (δ; posterior slope angle of the tibial component).
Rang of motion | 1 year
  Functional evaluation:it is measured by a blinded observer using goniometer.
patellar displacement (PD) | 1 year
  The patellar displacement is the lateral displacement of the median ridge of the patella from the intercondylar sulcus of the femur.The PD was assessed by a blinded observer using 30° skyline radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kuo Yu, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Abdel MP, Parratte S, Budhiparama NC. The patella in total knee arthroplasty: to resurface or not is the question. Curr Rev Musculoskelet Med. 2014 Jun;7(2):117-24. doi: 10.1007/s12178-014-9212-4. PMID 24706154
- [Background] Breeman S, Campbell M, Dakin H, Fiddian N, Fitzpatrick R, Grant A, Gray A, Johnston L, Maclennan G, Morris R, Murray D; KAT Trial Group. Patellar resurfacing in total knee replacement: five-year clinical and economic results of a large randomized controlled trial. J Bone Joint Surg Am. 2011 Aug 17;93(16):1473-81. doi: 10.2106/JBJS.J.00725. PMID 22204002
- [Background] Camp CL, Bryan AJ, Walker JA, Trousdale RT. Surgical technique for symmetric patellar resurfacing during total knee arthroplasty. J Knee Surg. 2013 Aug;26(4):281-4. doi: 10.1055/s-0032-1330056. Epub 2013 Jan 8. PMID 23299953
- [Background] Bartlett DH, Franzen J. Accurate preparation of the patella during total knee arthroplasty. J Arthroplasty. 1993 Feb;8(1):75-82. doi: 10.1016/s0883-5403(06)80111-7. PMID 8436994
- [Derived] Yuan F, Sun Z, Wang H, Chen Y, Yu J. Clinical and radiologic outcomes of two patellar resection techniques during total knee arthroplasty: a prospective randomized controlled study. Int Orthop. 2019 Oct;43(10):2293-2301. doi: 10.1007/s00264-018-4264-5. Epub 2018 Dec 11. PMID 30539221